CLINICAL TRIAL: NCT05589753
Title: Targeting Chemoreceptor Control of Breathing During Sleep to Mitigate Opioid-Associated Sleep Disordered Breathing
Brief Title: Sleep Disordered Breathing With Opioid Use
Acronym: SDB
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: John D. Dingell VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PULM-003-18F; 1904002203 (Other Grant/Funding Number: John D. Dingell VA Medical Center)
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Sleep Apnea; Opioid Use; Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Oxygen; Acetazolamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperoxia (Experimental): Determine the effect of sustained hyperoxia overnight vs room air overnight on ventilatory control during sleep, including the apneic threshold, carbon-dioxide reserve and chemosensitivity measured via pressure support ventilation (PSV) during non-rapid eye movement sleep (NREM) sleep.
  Interventions: Other: Hyperoxia
- Acetazolamide (ACZ) (Experimental): Determine the effect of acetazolamide on cerebrovascular responsiveness to CO2 during wake and sleep. Participants will receive oral ACZ therapy for 6 days, While on the medication following studies will be performed - experimental night study, experimental day study, polysomnography night study (PSG).
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Other: Hyperoxia — The ventilatory effects of brief hyperoxia will be assessed by analyzing control breaths on room air immediately preceding the hyperoxic exposure, and comparing with the primary end-point, nadir minute ventilation breath, immediately following the brief hyperoxic exposure.
  Other Names: oxygen
  Arms: Hyperoxia
Drug: Acetazolamide — Participants with sleep apnea will ingest capsules containing either placebo or acetazolamide 500 mg twice a day for 6 days. On the final 4 consecutive nights while still on ACZ, the investigators will perform i) physiology tests and ii) in-lab follow-up PSG.
  Other Names: ACZ
  Arms: Acetazolamide (ACZ)

SUMMARY:
There is an increased risk for sleep disordered breathing (SDB), sleep-related hypoventilation and irregular breathing in individuals on chronic prescription opioid medications. Almost 30% of a veteran sleep clinic population had opioid-associated central sleep apnea (CSA). The proposal aims to identity whether oxygen and acetazolamide can be effective in reducing unstable breathing and eliminating sleep apnea in chronic opioid use via different mechanisms. We will study additional clinical parameters like quality of life, sleep and pain in patients with and without opioid use. This proposal will enhance the investigators' understanding of the pathways that contribute to the development of sleep apnea with opioid use. The investigators expect that the results obtained from this study will positively impact the health of Veterans by identifying new treatment modalities for sleep apnea.

DETAILED DESCRIPTION:
In a national sample of Veterans, SDB was a significant risk factor for opioid-related toxicity and overdose; and the presence of CSA combined with chronic prescription opioid use compounded the mortality risk. There are only limited and partially effective therapies for this sleep disorder and the exact mechanisms by which opioids produce SDB in adults remain unclear, and varied and conflicting ventilatory control mechanisms have been suggested. This proposal will investigate whether alternative therapies can be developed by modulating specific physiologic mechanisms of ventilatory control. Specifically, the investigators will study effects of chronic oral prescription opioids on chemoresponsiveness and cerebrovascular responsiveness (CVR) (Aim 1); and whether interventions with sustained hyperoxia (Aim 2) and acetazolamide (Aim 3) will reduce the apneic threshold (AT) to alleviate breathing instability and SDB in chronic prescription opioid-associated SDB. The proposed aims will also allow us to delineate key mechanisms of breathing instability with opioid and without opioid use. The information garnered from the proposed experiments will drive development of novel personalized therapies to reduce SDB associated with chronic opioids in Veterans and, ultimately, will positively impact their long-term health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Veterans, age 18-89 years
* Veterans with prescription opioids

Exclusion Criteria:

* Patients with BMI>40kg/m2 will be excluded to avoid the effects of morbid obesity on pulmonary mechanics and ventilatory control
* Patients with history of unresolved/untreated cardiac disease, including recent myocardial infarction, recent bypass surgery, untreated atrial and ventricular tachy-bradycardias
* Congestive heart failure with Cheyne-Stokes respiration (CSR)
* Current unstable angina
* Recent stroke
* Untreated schizophrenia
* Untreated hypothyroidism
* Unresolved seizure disorder
* Severe respiratory, neurological, liver and renal diseases
* Unstable psychiatric disorders/untreated PTSD
* Traumatic brain injury
* Pregnant women
* Significant sleep disorder such as narcolepsy, parasomnias disorder
* Failure to give informed consent
* Patients on tramadol and suboxone/buprenorphine

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Apneic threshold- a measure of breathing instability | 2 days to 30 days
  Measures of breathing instability including: Apneic threshold: this is the end-tidal Co2 at which a central apnea closes to a hypopnea is produced.
Cerebrovascular responsiveness to carbon-dioxide | 7 days
  Cerebrovascular response to different levels of CO2: this is a measure of the response of the cerebral blood flow to changes in carbon dioxide levels and is used as a measure of ventilatory control of breathing
Ventilatory responsiveness | 2 days to 30 days
  Hypocapnic ventilatory response; this is calculated as the change in minute ventilation for corresponding changes in PETCO2.
Carbon -dioxide reserve | 2 days to 30 days
  This is a derived measure. This is calculated as the difference between the apneic threshold PETCO2 (given above) and the control PETCO2.

SECONDARY OUTCOMES:
Apnea hypopnea index | 2 days to 30 days
  Apnea hypopnea index- is a measure of severity of sleep apnea - this is calculated as the total number of apneas and hypopneas recorded during a sleep study divided by the total sleep time during the sleep study.

CONTACTS AND LOCATIONS:
Overall Officials: Susmita Chowdhuri, MD MS, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No